CLINICAL TRIAL: NCT02595060
Title: GM-CSF Inhalation to Improve Host Defense and Pulmonary Barrier Restoration (GI-HOPE). A Randomized, Double-blind, Parallel Group, Multicenter, Phase II Study
Brief Title: Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF) Inhalation to Improve Host Defense and Pulmonary Barrier Restoration
Acronym: GI-HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOL-ARDS-002
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: ARDS
Keywords: acute lung injury, molgramostim, GM-CSF, pneumonia, barrier restoration
MeSH Terms: conditions — Acute Lung Injury; Pneumonia | interventions — regramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 150 mcg inhaled molgramostim (Experimental): once daily inhaled molgramostim (rhGM-CSF) for 3 days
  Interventions: Drug: inhaled molgramostim (rhGM-CSF)
- 450 mcg inhaled molgramostim (Experimental): once daily inhaled molgramostim (rhGM-CSF) for 3 days
  Interventions: Drug: inhaled molgramostim (rhGM-CSF)
- inhaled placebo (Placebo Comparator): once daily inhaled placebo for 3 days
  Interventions: Drug: inhaled placebo

INTERVENTIONS:
Drug: inhaled molgramostim (rhGM-CSF)
  Arms: 150 mcg inhaled molgramostim; 450 mcg inhaled molgramostim
Drug: inhaled placebo — formulated as the active substance without molgramostim
  Arms: inhaled placebo

SUMMARY:
This trial evaluates efficacy and safety of inhaled molgramostim (rhGM-CSF) in 45 patients with pneumonia associated acute respiratory distress syndrome (ARDS). A third of the patients will receive 150 mcg inhaled molgramostim, another third 450 mcg and the remaining third will receive inhaled placebo for 3 days. The patients will be followed for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form by the patient or a legal representative according to local regulations
2. Man or woman 18 to 75 years of age, inclusive
3. Women who have been post-menopausal for more than 1 year or women of childbearing potential period using a highly efficient method of contraception (i.e. a method with less than 1% failure rate such as combined hormonal contraception, progesterone-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tube occlusion, vasectomized partner, sexual abstinence) during dosing and hospitalisation. Women must have a negative serum or urine pregnancy test before the first dose of study medication and must not be lactating.
4. Diagnosis of pneumonia-associated ARDS, where the underlying condition is Community-Acquired Pneumonia (CAP) or Hospital-Acquired Pneumonia (HAP) in patients not on invasive ventilation upon diagnosis of HAP.
5. Diagnosis of ARDS according to the Berlin ARDS definition.
6. Requirement for positive pressure ventilation (non-invasive or via endotracheal tube) for more than 72 hours in total with inspiratory oxygen concentration (FiO2) ≥ 50% (or less when on additional ECMO therapy) not longer than 14 days

Exclusion Criteria:

1. Receiving vasopressors of >100 µg/min
2. History of liver cirrhosis Child Pugh C, chronic hemodialysis (before severe pneumonia/ARDS), lung cancer
3. Malignancy with expected survival time of less than 6 months
4. History of or listing for lung transplantation
5. Highly immunosuppressive therapy or anti-malignant combination chemotherapy within 3 weeks prior to first dose of study drug
6. Any anti-malignant chemotherapy within 24 hours prior to first dose of study drug
7. AIDS or known history of HIV infection
8. Pregnancy
9. Autoimmune thrombocytopenia, myelodysplastic syndromes with > 20% marrow blast cells
10. History or presence of hypersensitivity or idiosyncratic reaction to molgramostim or to related compounds (i.e., Growgen®, Leucomax®, Leukine™, Topleucon™)
11. Participation in another clinical trial within 90 days prior to the first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
GI-HOPE score representing changes at Day 4/5 with respect to Baseline (Day -1) | baseline and Day 4/5
  The GI-HOPE score assesses change in bronchoalveolar lavage fluid (BALF) mononuclear phagocyte activation/polarization by flow cytometry (mean fluorescence intensities of parameters CD80, CD86, CD206, HLA-DR) with respect to baseline.

SECONDARY OUTCOMES:
Number of patients with Adverse Events (AE), Serious AEs and Adverse Drug Reactions | baseline to 28 days
Oxygenation | Baseline to Day 11
  PaO2/FiO2
Acute Physiology and Chronic Health Evaluation (APACHE) | Baseline to Day 11
Sequential Organ Failure Assessment (SOFA) | Baseline to Day 11
Extravascular Lung Water Index | Baseline to Day 11
C-reactive Protein | Baseline to Day 11
Days on vasoactive drugs | Baseline to Day 28
All cause mortality | Baseline to Day 28
Serum GM-CSF | Baseline, Days 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Herold, Prof.Dr.med.,PhD, Principal Investigator — Universities of Giessen and Marburg Lung Centers, Germany
Locations (7):
- Germany (7):
  - Klinik und Poliklinik für Anästhesiologie, Intensivmedizin, Notfallmedizin und Schmerztherapie, Würzburg, Baden-Würtemberg
  - Universitätsklinikum Frankfurt, Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Frankfurt
  - Universities of Marburg and Giessen Lung Center, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Intensivmedizin, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Pneumologie, Hanover
  - Universitätsklinikum Jena, Klinik für Anästhesiologie und Intensivmedizin, Jena
  - University Hospital Marburg, Department of Anaesthesiology and Intensive Care Medicine, Marburg

REFERENCES:
- [Background] Herold S, Hoegner K, Vadasz I, Gessler T, Wilhelm J, Mayer K, Morty RE, Walmrath HD, Seeger W, Lohmeyer J. Inhaled granulocyte/macrophage colony-stimulating factor as treatment of pneumonia-associated acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Mar 1;189(5):609-11. doi: 10.1164/rccm.201311-2041LE. No abstract available. PMID 24579839
- [Background] Cakarova L, Marsh LM, Wilhelm J, Mayer K, Grimminger F, Seeger W, Lohmeyer J, Herold S. Macrophage tumor necrosis factor-alpha induces epithelial expression of granulocyte-macrophage colony-stimulating factor: impact on alveolar epithelial repair. Am J Respir Crit Care Med. 2009 Sep 15;180(6):521-32. doi: 10.1164/rccm.200812-1837OC. Epub 2009 Jul 9. PMID 19590023
- [Background] Unkel B, Hoegner K, Clausen BE, Lewe-Schlosser P, Bodner J, Gattenloehner S, Janssen H, Seeger W, Lohmeyer J, Herold S. Alveolar epithelial cells orchestrate DC function in murine viral pneumonia. J Clin Invest. 2012 Oct;122(10):3652-64. doi: 10.1172/JCI62139. Epub 2012 Sep 10. PMID 22996662
- [Background] Ballinger MN, Paine R 3rd, Serezani CH, Aronoff DM, Choi ES, Standiford TJ, Toews GB, Moore BB. Role of granulocyte macrophage colony-stimulating factor during gram-negative lung infection with Pseudomonas aeruginosa. Am J Respir Cell Mol Biol. 2006 Jun;34(6):766-74. doi: 10.1165/rcmb.2005-0246OC. Epub 2006 Feb 10. PMID 16474098
- [Background] Standiford LR, Standiford TJ, Newstead MJ, Zeng X, Ballinger MN, Kovach MA, Reka AK, Bhan U. TLR4-dependent GM-CSF protects against lung injury in Gram-negative bacterial pneumonia. Am J Physiol Lung Cell Mol Physiol. 2012 Mar 1;302(5):L447-54. doi: 10.1152/ajplung.00415.2010. Epub 2011 Dec 9. PMID 22160309